CLINICAL TRIAL: NCT04012723
Title: Clinical Trial of a New Device for Real-Time Muscle Pressure Measurements in Patients With an Upper or Lower Extremity Fracture at Risk for Acute Compartment Syndrome
Brief Title: Clinical Trial of a New Device for Real-Time Muscle Pressure Measurements in Patients at Risk for Acute Compartment Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MY01 Inc. (Industry)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MY01-NS-01
Record Dates: First submitted 2019-07-03; First posted 2019-07-09 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Compartment Syndrome Traumatic Lower Extremity; Compartment Syndrome Traumatic Upper Extremity
Keywords: Acute Compartment Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MY01 Device (Experimental): Device: MY01 Device
  Insertion of the MY01 device for up to 24 hours for continuous monitoring of compartment pressure
  Interventions: Device: MY01 Continuous Compartmental Pressure Monitor

INTERVENTIONS:
Device: MY01 Continuous Compartmental Pressure Monitor — The MY01 Continuous Compartmental Pressure Monitor is intended for real-time and continuous measurement of compartmental pressures.

SUMMARY:
Compartment syndrome remains a very serious complication of lower extremity trauma and/or procedural cases that involved lower or upper extremity surgery. This condition results in muscle death, chronic pain, infection, and possible amputation. Early diagnosis is essential to institute interventions to avoid complications. Unfortunately, the subjective pain of the patient remains the mainstay for diagnosis. A method or device is needed that would improve the investigator's ability to diagnose this potentially devastating condition. The purpose of this trial is to evaluate the safety and functionality of MY01, an investigational device that allows continuous monitoring of intracompartmental muscle pressure in patients at risk for developing acute compartment syndrome. This is a single centre, non-randomized, non-controlled, unblinded, prospective trial of the MY01 device. A cohort of 25 participants will be prospectively enrolled to document the performance of the device.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 16-65.
* Fracture of the tibia, foot, forearm, femur, or humerus that is felt by the surgeon to have a reasonable indication that elevated intracompartmental pressure could occur in the patient.
* Planned admission to hospital (to enable monitoring of compartment pressures)
* Provision of informed consent to participate.

Exclusion Criteria:

* Frankly contaminated or infected wounds or fractures.
* Clinical suspicion of acute compartment syndrome requiring urgent fasciotomy at time of presentation to study center.
* Current or pre-existing neuropathy in the study limb.
* Pregnant women.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Clinical ease with which the MY01 device is able to be inserted into a compartment. | 24-48 hours following device insertion.
  At device insertion, the physician will complete a feedback questionnaire, and routine assessment will be performed in compliance with the standard of care. As part of the feedback questionnaire, the physician will be asked to indicate on a sliding scale "How certain are you that the sensor is in the correction position?" [1 = uncertain] - [5 = very certain].
  The scale, administered part of a Clinical Report Form (CRF) titled 'Physician Survey', measures the physicians subjective level of certainty that the device sensor was inserted correctly within a patients muscle compartment. A record of 5 should be considered a positive scenario, whereas a record of 1 should indicate a negative scenario.
Ability to monitor in real time the continuous pressure readout from the compartment in remote locations via smartphone. | 24-48 hours following device insertion.
  At insertion of device the physician will complete a feedback questionnaire on the device, the participant will be assessed for adverse events, and routine assessment will be performed.
The change in intracompartmental pressure. | 24-48 hours following device insertion.
  Routine assessments will be completed by healthcare personnel as per standard of care (the 6P's [Pain, Paraesthesia, Pallor, Paralysis, Pulselessness, Poikilothermia]), and compared against the pressure readout [mmHG] indicated by MY01's MicroElectroMechanical (MEMS) pressure sensor inserted at the afflicted location.

SECONDARY OUTCOMES:
Adverse events associated with the use of the device. | 24-48 hours following device insertion, and again during the final follow-up of the participant approximately two weeks after treatment.
  The patient will be monitored for adverse events during treatment, and will be reassessed during the final follow-up of the participant at the first return visit to the fracture clinic. An adverse event constitutes "Any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal lab findings) in participants, users or other persons, whether or not related to the investigational device."
Pain at insertion site. | 24-48 hours following device insertion.
  Participants will be asked to keep a diary while the device is in situ. The diary will consist of a pain Visual Analog Score (VAS) to be completed each time their vitals are taken, with space to freely comment on the device. VAS will be on a sliding scale where [0=no pain] and [10=pain as bad as it can be].

CONTACTS AND LOCATIONS:
Overall Officials: Ross Leighton, MD, Principal Investigator — Orthopaedic Surgeon, Nova Scotia Health Authority
Locations (5):
- Canada (5):
  - Foothills Medical Center, Calgary, Alberta
  - Halifax Infirmary, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - Ottawa Civic Hospital, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No